CLINICAL TRIAL: NCT06079918
Title: Individually Randomized Trial of Higher-dose Iron (60 mg, 45 mg) Compared to Low-dose Iron (30 mg) in Multiple Micronutrient Supplements in Pregnancy on Moderate and Severe Maternal Anemia
Brief Title: Multiple Micronutrient Supplementation for Maternal Anemia Prevention in Tanzania
Acronym: MMS-MAP
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: George Washington University (Other)
Collaborators: Ifakara Health Institute (Other); Harvard School of Public Health (HSPH) (Other); Muhimbili University of Health and Allied Sciences (Other); Africa Academy for Public Health (Other); Columbia University (Other)
Responsible Party: Principal Investigator, Emily Smith, Principal Investigator, George Washington University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MMS-MAP
Record Dates: First submitted 2023-07-25; First posted 2023-10-12 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Pregnancy Related
Keywords: Pregnancy; Multiple Micronutrient Supplementation; Iron; Anemia; Tanzania
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The trial is quadruple blind with all trial participants, outcome assessors (research staff and care providers), investigators, and trials statistician and data analysts being unable to determine the allocated trial arm for any trial participant or identify trial participants who are on the same trial regimen.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- MMS with 30 mg iron (Active Comparator): MMS with standard UNIMMAP formulation of 15 micronutrients, including 30 mg of iron
  Interventions: Dietary Supplement: Multiple Micronutrient Supplements with 30 mg of elemental iron
- MMS with 45 mg iron (Experimental): MMS with 45 mg of iron plus standard UNIMMAP formulation for other 14 micronutrients
  Interventions: Dietary Supplement: Multiple Micronutrient Supplements with 45 mg of elemental iron
- MMS with 60 mg iron (Experimental): MMS with 60 mg of iron plus standard UNIMMAP formulation for other 14 micronutrients
  Interventions: Dietary Supplement: Multiple Micronutrient Supplements with 60 mg of elemental iron

INTERVENTIONS:
Dietary Supplement: Multiple Micronutrient Supplements with 30 mg of elemental iron — MMS with 30 mg iron is the active comparator group. The standard UNIMMAP MMS formulation includes 30 mg of iron which will be taken orally once daily from the time of randomization until delivery.
  Arms: MMS with 30 mg iron
Dietary Supplement: Multiple Micronutrient Supplements with 45 mg of elemental iron — MMS with 45 mg iron is an intervention group. MMS with 45 mg of iron plus standard UNIMMAP formulation for other 14 micronutrients will be taken orally once daily from the time of randomization until delivery.
  Arms: MMS with 45 mg iron
Dietary Supplement: Multiple Micronutrient Supplements with 60 mg of elemental iron — MMS with 60 mg iron is an intervention group. MMS with 60 mg of iron plus standard UNIMMAP formulation for other 14 micronutrients will be taken orally once daily from the time of randomization until delivery.
  Arms: MMS with 60 mg iron

SUMMARY:
This is an individually randomized controlled trial to assess the effect of multiple micronutrient supplements (MMS) containing 60 and 45 mg iron as compared to MMS containing 30 mg of iron (standard UNIMMAP formulation) on maternal moderate or severe anemia. This study will help inform countries like Tanzania that currently use IFA containing 60 mg of iron regarding the dose of iron to use in MMS.

ELIGIBILITY:
Inclusion Criteria:

* Attending first ANC visit at study clinics
* Pregnant women < 20 weeks gestation by last menstrual period (LMP)
* Aged ≥ 18 years old
* Intending to stay in Dar es Salaam until 6 weeks post delivery
* Provides informed consent

Exclusion Criteria:

* Severe anemia (defined as hemoglobin < 8.5 g/dL per Tanzania standard of care)
* Sickle cell disease (SS and SC) and hemoglobin C disease (CC) as tested by HemoTypeSC
* Concurrently enrolled in another nutritional clinical trial
* Pregnant women with disability or condition which would impair their ability to provide informed consent and complete study procedures.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6381 (Estimated)
Dates: Start 2025-03-03 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Proportion of pregnant women with third-trimester moderate or severe anemia | 3rd trimester (weeks 28-42 of pregnancy)
  Defined as a hemoglobin concentration <10 g/dL.

SECONDARY OUTCOMES:
Maternal hemoglobin concentration | 3rd trimester (weeks 28-42 of pregnancy)
  Continuous hemoglobin concentration measured from venous blood by complete blood count
Maternal hemoglobin concentration | 6 weeks postpartum
  Continuous hemoglobin concentration measured from venous blood by complete blood count
Proportion of pregnant women with anemia | 3rd trimester (weeks 28-42 of pregnancy)
  Hb concentration < 11 g/dL
Proportion of postpartum women with anemia | 6 weeks postpartum
  Hb concentration < 12 g/dL
Maternal serum ferritin | 3rd trimester (weeks 28-42 of pregnancy)
  Inflammation-adjusted serum ferritin
Proportion of pregnant women with iron deficiency | 3rd trimester (weeks 28-42 of pregnancy)
  Inflammation-adjusted serum ferritin < 15 ug/L
Proportion of pregnant women with iron deficiency anemia | 3rd trimester (weeks 28-42 of pregnancy)
  Anemia (Hb < 11 g/dL) and iron deficiency (inflammation-adjusted serum ferritin < 15 ug/L)
Proportion of women with preeclampsia | From 20 weeks gestation through delivery
  Gestational hypertension and gestational proteinuria among participants without chronic hypertension or gestational proteinuria among participants with chronic hypertension (superimposed preeclampsia) or clinical diagnosis of preeclampsia by managing clinical team or development of severe features of preeclampsia even in the absence of proteinuria
Proportion of women with antepartum bleeding | From 24 weeks gestation through delivery
  Self-reported or clinical diagnosis of bleeding from or into the genital tract
Proportion of women with postpartum hemorrhage | From delivery through 42 days post delivery
  Clinical diagnosis of postpartum hemorrhage or use of critical interventions to treat postpartum hemorrhage
Proportion of women with infection-related severe maternal outcomes | During pregnancy through 42 days postpartum
  Severe infection-related such as hospitalization for infection, women presenting with WHO near-miss criteria to define organ system dysfunction, invasive procedure to treat the source of infection (vacuum aspiration, dilatation and curettage, wound debridement, drainage, laparotomy and lavage, other surgery), or maternal death from infection.
Proportion of women with pregnancy-related death | Pregnancy through 42 days of pregnancy termination
  Death of a woman while pregnant or within 42 days of termination of pregnancy, irrespective of the cause of death
Proportion of women with symptoms consistent with depression | 3rd trimester (weeks 28-42 of pregnancy)
  Patient Health Questionnaire-9 (PHQ-9) score ranging from 0 to 27, with higher scores consistent with depression and anxiety
Proportion of women with symptoms consistent with depression | 6 weeks postpartum
  Patient Health Questionnaire-9 (PHQ-9) score ranging from 0 to 27, with higher scores consistent with depression and anxiety
Proportion of women with symptoms consistent with fatigue | 3rd trimester (weeks 28-42 of pregnancy)
  FACIT assessment score ranging from 0 to 52, with lower scores consistent with fatigue.
Proportion of women with symptoms consistent with fatigue | 6 weeks postpartum
  FACIT assessment score ranging from 0 to 52, with lower scores consistent with fatigue.
Proportion of women with malaria infection | Pregnancy through 42 days postpartum
  Based on HRP2 biomarker or rapid-diagnostic tests (RDTs)
Proportion of fetal deaths | At pregnancy termination (weeks 1-42 of pregnancy)
  A product of human conception, irrespective of the duration of the pregnancy, which, after expulsion or extraction, does not breath or show any other evidence of life such as beating of the heart, pulsation of the umbilical cord, or definite movement of voluntary muscles, whether or not the umbilical cord has been cut or the placenta is attached
Proportion of stillbirths | At pregnancy termination (weeks 1-42 of pregnancy)
  Fetal death ≥ 28 weeks gestation
Birthweight | At birth
  Continuous birthweight among live births
Proportion of live births with low birthweight | At birth
  Live birth with birthweight < 2500 g
Gestational age at birth | At birth
  Duration of gestation in weeks as a continuous measure among live births based on best obstetric estimate among live births
Proportion of preterm live births | At birth
  Live birth <37 weeks gestation (based on best obstetric estimate)
Birthweight for gestational age | At birth
  Continuous centile based on INTERGROWTH-21st standard birth centile among live births
Proportion of small-for-gestational age live births (<10th percentile) | At birth
  Size-for-gestational age <10th on the INTERGROWTH-21st standard among live births
Proportion of small-for-gestational age live births (<3rd percentile) | At birth
  Size-for-gestational age <3rd percentile on the INTERGROWTH-21st standard among live births
Infant hemoglobin concentration | At 6 weeks of age
  Continuous Hb concentration measured from capillary blood by complete blood count
Infant serum ferritin | At 6 weeks of age
  Continuous inflammation adjusted serum ferritin
Proportion of infants with iron deficiency | At 6 weeks of age
  Inflammation-adjusted serum ferritin < 20 ug/L
Proportion of neonatal deaths | From birth to 28 days of age
  Death of liveborn infant during the first 28 completed days of life
Proportion of infant deaths < 42 days | From birth to 42 days of age
  Death of a live born infant during the first 42 completed days of life

OTHER OUTCOMES:
Percent adherence | During pregnancy (up to week 42)
  The percentage of days a pregnant woman takes a MMS pill out of the total number of days from randomization to delivery
Diarrhea | During pregnancy (up to week 42)
  Self-reported any diarrhea symptoms during the intervention period
Heartburn | During pregnancy (up to week 42)
  Self-reported any heartburn symptoms during the intervention period
Constipation | During pregnancy (up to week 42)
  Self-reported any constipation symptoms during the intervention period
Vomiting | During pregnancy (up to week 42)
  Self-reported any vomiting symptoms during the intervention period
Nausea | During pregnancy (up to week 42)
  Self-reported any nausea symptoms during the intervention period
Leg Cramps | During pregnancy (up to week 42)
  Self-reported any leg cramps during the intervention period
Low back/pelvic pain | During pregnancy (up to week 42)
  Self-reported any low back/pelvic pain during the intervention period
Maternal blood lead concentration | 3rd trimester (weeks 28-42 of pregnancy)
  Continuous blood lead concentration measured from whole blood
Maternal plasma zinc concentration | 3rd trimester (weeks 28-42 of pregnancy)
  Continuous zinc concentration measured from plasma

CONTACTS AND LOCATIONS:
Overall Officials: Blair Wylie, MD, MPH, Principal Investigator — Columbia University; Honorati Masanja, PhD, Principal Investigator — Ifakara Health Institute; Alfa Muhihi, MD, MPH, Principal Investigator — Africa Academy for Public Health; Andrea Pembe, MD, MMed, PhD, FCOG, Principal Investigator — Muhimbili University of Health and Allied Sciences; Emily R Smith, ScD, MPH, Principal Investigator — The Goerge Washington University; Christopher R Sudfeld, ScD, ScM, Principal Investigator — Harvard University
Locations (1):
- Muhimbili University of Health and Allied Sciences, Dar es Salaam, Tanzania

REFERENCES:
- [Derived] Smith ER, Muhihi A, Wylie BJ, Mugusi S, Aboud S, Bakari M, Fawzi W, Kinyogoli S, Oakley EM, Pan Q, Sando MM, Brownlee VS, Pembe AB, Sudfeld CR, Masanja H. Multiple micronutrient supplementation for maternal anemia prevention (MMS-MAP): an individually randomized trial of higher-dose iron (60 mg, 45 mg) compared to low-dose iron (30 mg) in multiple micronutrient supplements in pregnancy. Trials. 2025 Jun 14;26(1):206. doi: 10.1186/s13063-025-08906-7. PMID 40517226